CLINICAL TRIAL: NCT06774456
Title: Validation of a 3D Motion Analysis Protocol With an Instrumented Game to Evaluate Upper Limb Impairments in Children With Neuromotor Disorders
Brief Title: Validation of a 3D Instrumented Serious Game to Evaluate Upper Limb Impairments in Children With Neuromotor Disorders
Acronym: Play2BEAPI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Marine Cacioppo, MD, PhD, University Hospital, Geneva
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-02423
Record Dates: First submitted 2025-01-02; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Cerebral Palsy; Brain Injury; Neurological; Disorder, Nervous System
Keywords: Children; upper limb; motion analysis; serious game; neuromotor disorders; bimanual function; electromyography
MeSH Terms: conditions — Cerebral Palsy; Brain Injuries; Neurologic Manifestations | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children with neuromotor disorders (Other): During Visit 1, children will perform both a validated 3D protocol and the instrumented 3D serious game (developed version). After each session, questionnaires will be distributed to participants to assess the added value of the immersive environment.
  During Visit 2, children will have a clinical examination (goniometry, muscle strength, spasticity, motor selectivity) and functional assessments by experienced therapists at hospital and will perform the instrumented 3D serious game.
  Interventions: Device: instrumented 3D serious game (BE API 3.0)
- Typically developing children (Other): Children will have one visit to the hospital (Visit 1). They will perform the instrumented serious game, in order to assess the discriminant validity of the upper limb movement features between children with neuromotor disorders and typically developing children.
  Interventions: Device: instrumented 3D serious game (BE API 3.0)

INTERVENTIONS:
Device: instrumented 3D serious game (BE API 3.0) — It is composed of bimanual tasks integrated into a game scenario. The child is first equipped with markers on the upper limb (UL) and trunk (3D motion analysis and electromyography), and he/she can then play the game. There are several tasks ('piloting missions') to evaluate specific UL movements. The UL movements are recorded when the child is playing. The instruments of the set-up (wheel, turbo, etc.) are connected to the game to play and can also be used as measurements (grip strength, etc.). The markers are then removed. The total duration of the game is about 30-45 minutes, including placing/removing markers and the game.
  Other Names: Clinical and functional tests; Validated 3D protocol (old version); Questionnaires

SUMMARY:
The goal of this clinical trial is to validate an instrumented 3D serious game to assess upper limb impairments in children with neuromotor disorders. The main questions are:

* Does an instrumented 3D serious game can provide a set of validated upper limb movement features with good reliability, validity and responsiveness ?
* Does the instrumented 3D serious game could provide better immersion, adhesion, usability and satisfaction than a "classic" 3D protocol, thanks to the developped environment ?

Researchers will compare children with neuromotor disorders and typically developing children to assess discriminant validity of the new assessement.

Children with neuromotor disorders will have 2 visits to the hospital :

* Visit 1 : children will perform a validated 3D protocol and the instrumented 3D serious game
* Visit 2 : children will have a clinical examination and will perform the instrumented 3D serious game

Typically developing children will have one visit to the hospital. They will perform the instrumented 3D serious game.

DETAILED DESCRIPTION:
The instrumented 3D serious game (BE API 3.0) will be performed during a 3D motion analysis session. It is composed of:

* One screen (35 pouces)
* Game set up (2-handed joystick, turbo, shifter, dashboard, box, coins and buzzer) instrumented with sensors to link the game and measure grasp strength.
* Software: Unity software (version 2022.3.21f1, Unity Technologies, San Francisco, California, USA)

The game is composed of bimanual tasks integrated into a game scenario. The child is first equipped with markers on the UL and trunk, and he/she can then play the game. There are several tasks ('piloting missions') to evaluate specific UL movements. The UL movements are recorded when the child is playing. The instruments of the set-up (wheel, turbo, etc.) are connected to the game to play and can also be used as measurements (grip strength, etc.). The markers are then removed. The total duration of the game is about 30-45 minutes, including placing/removing markers and the game.

ELIGIBILITY:
Inclusion Criteria:

* Children with NMD

  * Informed Consent signed by the subject
  * Aged from 5 to 13 years,
  * Non-progressive neurological lesions (cerebral palsy, stroke, traumatic brain injury, etc.),
  * With sufficient grasp ability to perform the 3D protocol tasks (MACS level I to III),
* TD children

  * Informed Consent signed by the subject
  * Aged from 5 to 13 years,

Exclusion Criteria:

* Children with neuromotor disorders

  * inability to follow the procedures of the investigation because of severe cognitive or visual disturbances,
  * upper limb (UL) disorders that may affect movement (fractures less than 6 months prior to participation, pain (visual analogic score (VAS) score > 0), etc.).
  * previous UL surgery, and botulinum toxin injections less than three months prior to participation,
* TD children

  * Inability to follow the procedures of the investigation because of severe visual disturbances,
  * UL disorders that may affect movement (fractures less than 6 months prior to participation, pain (VAS score > 0), etc.).

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Arm Profile Score | Baseline and 2 weeks after
  A kinematic index (upper limb movement feature) which reflects the severity of the deviations of the subject's movement compared with a group of typically developing children. The measure ranges from 0° to infinity. The measure is expressed in degrees. The higher the measure, the more abnormal the deviation is.

SECONDARY OUTCOMES:
Kinematics | Baseline and 2 weeks after
  Joint angular values, in degrees
Movement quality - smoothness | Baseline and 2 weeks after
  A movement features obtained with 3D motion analysis (spectral arc length). No unit
Movement quality - trajectory | Baseline and 2 weeks after
  A movement features obtained with 3D motion analysis (index of curvature), in degrees
Spatiotemporal - velocity | Baseline and 2 weeks after
  A movement features obtained with 3D motion analysis. Velocity, in meter/seconds
Spatiotemporal - duration | Baseline and 2 weeks after
  A movement features obtained with 3D motion analysis. Duration in seconds
Electromyography | Baseline and 2 weeks after
  muscle activity in microVolt
Muscle strength | 1 day
  Muscle strength will be evaluated using the Medical Research Council scale (Paternostro-Sluga et al., 2008), a six-point ordinal scale from 0 to 5 in which 0 indicates no muscle contraction and 5 indicates normal strength. A composite strength score will be defined as the sum of the muscle weakness scores (total score: 0-80).
Muscle spasticity | 1 day
  Muscle spasticity will be evaluated with the Modified Ashworth Scale (MAS) (Mutlu et al., 2008), a six-point ordinal scale, rating from 0 to 4 (possible scores: 0,1,1+,2,3,4). A score of 0 represents normal muscle tone, whereas a score of 4 corresponds to no possible movement due to rigidity. A composite spasticity score, rated from 0 to 5, will be defined as the sum of MAS scores for each child (total score: 0-80 [16 muscles × 5 levels]).
Muscle selectivity | 1 day
  Muscle selectivity was evaluated using selective motor control (SMC) (Masson, n.d.), a five-point ordinal scale from 0 to 2, in increments of 0.5, in which a score of 2 corresponded to normal selectivity. A composite selectivity score was defined as the sum of the muscle selectivity scores (total score: 0-32).
Melbourne Assessment Test | 1 day
  It is a valid and reliable criterion-referenced test of impaired upper limb movement quality. The final score is reported as 4 separate sub-scores, 1 for each item of movement quality, reported on a scale from 0-100%, where 100% corresponds to full functional capacity.
Assisting Hand Assessment (AHA) | 1 day
  It is video recorded and rated using video-based scoring. It involves the evaluation of 22 bimanual activities. The total score ranges from 0 to 100 AHA-units; 100 AHA-units indicates normal spontaneous use of the impaired hand.
Abilhand-Kids | 1 day
  It is a questionnaire of bimanual daily life activities addressed to parents. Parents are asked to rate their child's difficulty on a 3-level scale (range from 0 to 2) for 21 items. The manual ability scale is calibrated in logits (i.e., log-odds units).
Short Feedback Questionnaire | 1 day
  It is a short post-immersive and presence questionnaire containing only six questions. Each item is rated from 0 to 5 (1 = not at all ; 5 = very much)
User Satisfaction Evaluation Questionnaire | 1 day
  It is a questionnaire developed in order to evaluate user satisfaction with rehabilitation systems. It comprises six questions that can be rated on a Likert scale ranging from 1 (not at all) to 5 (very much).
System Usability Scale | 1 day
  It is a questionnaire of usability. It is composed of 10 items. Only for the purpose of this study, the word "interface" in the items has been used interchangeably with the word "game". Each item's score ranged from 0 to 4. For items 1, 3, 5, 7 and 9 (odd-numbered items) the score contribution was the scale position minus 1. For items 2, 4, 6, 8 and 10 (even-numbered items) the score contribution was 5 minus the scale position. Next, we multiplied the sum of scores by 2.5 to obtain the overall System Usability value. SUS scores range from 0 to 100.

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospital, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cacioppo M, Loos A, Lempereur M, Brochard S. Bimanual movements in children with cerebral palsy: a systematic review of instrumented assessments. J Neuroeng Rehabil. 2023 Feb 27;20(1):26. doi: 10.1186/s12984-023-01150-7. PMID 36849971
- [Background] Gaillard F, Cacioppo M, Bouvier B, Bouzille G, Newman CJ, Pasquet T, Cretual A, Rauscent H, Bonan I. Assessment of bimanual performance in 3-D movement analysis: Validation of a new clinical protocol in children with unilateral cerebral palsy. Ann Phys Rehabil Med. 2020 Oct;63(5):408-415. doi: 10.1016/j.rehab.2019.06.008. Epub 2019 Jul 10. PMID 31301386
- [Background] Cacioppo M, Lempereur M, Houx L, Bouvier S, Bailly R, Brochard S. Detecting Movement Changes in Children with Hemiparesis after Upper Limb Therapies: A Responsiveness Analysis of a 3D Bimanual Protocol. Sensors (Basel). 2023 Apr 24;23(9):4235. doi: 10.3390/s23094235. PMID 37177439
- [Background] Cacioppo M, Marin A, Rauscent H, Le Pabic E, Gaillard F, Brochard S, Garlantezec R, Cretual A, Bonan I. A new child-friendly 3D bimanual protocol to assess upper limb movement in children with unilateral cerebral palsy: Development and validation. J Electromyogr Kinesiol. 2020 Dec;55:102481. doi: 10.1016/j.jelekin.2020.102481. Epub 2020 Oct 10. PMID 33091791